CLINICAL TRIAL: NCT02269735
Title: A Three-part Study Parts I, II and III: Rising Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of MK-2640 in Healthy Subjects (Part I) and Evaluation of Safety, Pharmacokinetics and Pharmacodynamics of MK-2640 in Subjects With Type 1 Diabetes Mellitus (Part II and Part III).
Brief Title: A Three-part Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of MK-2640 in Healthy Participants (Part I) and Participants With Type 1 Diabetes Mellitus (Parts II and III) (MK-2640-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2640-001
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — MK-2640; Insulin; Glucose; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- Part I: MK-2640 (Panel A) (Experimental): Part I: Lowest dose of MK-2640 infusion (3 approximately three-hour infusions at escalating rates) and dextrose infusion for 9 hours.
  Interventions: Drug: MK-2640; Drug: Dextrose; Drug: Rescue medication
- Part I: MK-2640 (Panel B) (Experimental): Part I: Low dose of MK-2640 infusion (3 approximately three-hour infusions at escalating rates) and dextrose infusion for 9 hours.
  Interventions: Drug: MK-2640; Drug: Dextrose; Drug: Rescue medication
- Part I: MK-2640 (Panel C) (Experimental): Part I: Medium-low dose of MK-2640 infusion (3 approximately three-hour infusions at escalating rates) and dextrose infusion for 9 hours.
  Interventions: Drug: MK-2640; Drug: Dextrose; Drug: Rescue medication
- Part I: MK-2640 (Panel D) (Experimental): Part I: Medium dose of MK-2640 infusion (3 approximately three-hour infusions at escalating rates) and dextrose infusion for 9 hours.
  Interventions: Drug: MK-2640; Drug: Dextrose; Drug: Rescue medication
- Part I: MK-2640 (Panel E) (Experimental): Part I: Medium-high dose of MK-2640 infusion (3 approximately three-hour infusions at escalating rates) and dextrose infusion for 9 hours.
  Interventions: Drug: MK-2640; Drug: Dextrose; Drug: Rescue medication
- Part I: MK-2640 (Panel F) (Experimental): Part I: High dose of MK-2640 infusion (3 approximately three-hour infusions at escalating rates) and dextrose infusion for 9 hours.
  Interventions: Drug: MK-2640; Drug: Dextrose; Drug: Rescue medication
- Part I: MK-2640 (Panel G) (Experimental): Part 1: Highest dose of MK-2640 infusion (3 approximately three-hour infusions at escalating rates) and dextrose infusion for 9 hours.
  Interventions: Drug: MK-2640; Drug: Dextrose; Drug: Rescue medication
- Part II: MK-2640 followed by RHI (Experimental): Part II: MK-2640 infusion and dextrose infusion for 9 hours during Period 1 of Part II followed by a 7-day wash-out period followed by RHI infusion and dextrose infusion for 9 hours during Period 2 of Part II. Insulin aspart administered approximately 10 hours before Periods 1 and 2 of Part II.
  Interventions: Drug: MK-2640; Biological: Regular Human Insulin (RHI); Drug: Dextrose; Biological: Insulin aspart; Drug: Rescue medication
- Part II: RHI followed by MK-2640 (Experimental): Part II: RHI infusion and dextrose infusion for 9 hours during Period 1 of Part II followed by a 7-day wash-out period followed by MK-2640 infusion and dextrose infusion for 9 hours during Period 2 of Part II. Insulin aspart administered approximately 10 hours before Periods 1 and 2 of Part II.
  Interventions: Drug: MK-2640; Biological: Regular Human Insulin (RHI); Drug: Dextrose; Biological: Insulin aspart; Drug: Rescue medication
- Part III: MK-2640 followed by RHI (Experimental): Part III: MK-2640 infusion and dextrose infusion for 7 hours during Period 1 of Part III followed by a 7-day wash-out period followed by RHI infusion and dextrose infusion for 7 hours during Period 2 of Part III. Insulin aspart administered approximately 10 hours before Periods 1 and 2 of Part III.
  Interventions: Drug: MK-2640; Biological: Regular Human Insulin (RHI); Drug: Dextrose; Biological: Insulin aspart; Drug: Rescue medication
- Part III: RHI followed by MK-2640 (Experimental): Part III: RHI infusion and dextrose infusion for 7 hours during Period 1 of Part III followed by a 7-day wash-out period followed by MK-2640 infusion and dextrose infusion for 7 hours during Period 2 of Part III. Insulin aspart administered approximately 10 hours before Periods 1 and 2 of Part III.
  Interventions: Drug: MK-2640; Biological: Regular Human Insulin (RHI); Drug: Dextrose; Biological: Insulin aspart; Drug: Rescue medication

INTERVENTIONS:
Drug: MK-2640 — MK-2640 intravenous infusion administered to participant in a fasted state
Biological: Regular Human Insulin (RHI) — RHI 100 units/mL intravenous infusion to maintain target glycemic level
  Arms: Part II: MK-2640 followed by RHI; Part II: RHI followed by MK-2640; Part III: MK-2640 followed by RHI; Part III: RHI followed by MK-2640
Drug: Dextrose — Dextrose 20% or 50% intravenous infusion for approximately 9 or 7 hours, as appropriate to attain a target glycemic level
Biological: Insulin aspart — Insulin aspart subcutaneous injection or intravenous infusion the evening before each period in Parts II and III to achieve/maintain glycemic target.
  Arms: Part II: MK-2640 followed by RHI; Part II: RHI followed by MK-2640; Part III: MK-2640 followed by RHI; Part III: RHI followed by MK-2640
Drug: Rescue medication — Rescue medication may be administered for hypotension or mild to moderate infusion reaction. Rescue medication may include epinephrine, antihistamines, steroids, or acetaminophen/paracetamol.

SUMMARY:
The purpose of Part I of this study is to evaluate the safety and tolerability of intravenous (IV) doses of MK-2640 in healthy participants and to obtain preliminary plasma pharmacokinetic profiles of MK-2640. The purpose of Parts II and III of this study is to evaluate the safety and tolerability of IV doses of MK-2640 and regular human insulin (RHI), and to evaluate the pharmacokinetic and pharmacodynamic profile of MK-2640 and RHI in participants with type 1 diabetes mellitus (T1DM). Part II will be initiated only if Part I general safety, tolerability and other observed data are supportive of progression to Part II. Part III will be initiated only if Parts I and II general safety, tolerability and other observed data are supportive of progression to Part III.

ELIGIBILITY:
Inclusion Criteria (Part I):

* healthy male or healthy female of non-child bearing potential
* in good health
* is a non-smoker and/or has not used nicotine or nicotine-containing products (e.g., nicotine patch) for at least approximately 3 months

Inclusion Criteria (Parts II and III):

* male or female of non-child bearing potential
* has T1DM for at least 12 months
* on stable doses of insulin
* in good health
* is a nonsmoker and/or has not used nicotine or nicotine-containing products (e.g., nicotine patch) for at least approximately 3 months

Exclusion Criteria:

* is mentally or legally incapacitated, or has significant emotional problems at the time of screening visit or expected during the conduct of the trial or has a history of clinically significant psychiatric disorder of the last 5 years
* has a history of clinically significant endocrine (except T1DM for Part II subjects), gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological (including stroke and chronic seizures) abnormalities or diseases
* is positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV)
* has a history of cancer (malignancy), except adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix
* has a history of significant multiple and/or severe allergies, or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food, had major surgery, donated or lost 1 unit of blood within 4 weeks prior to the screening visit
* has participated in another investigational trial within 4 weeks prior to the screening visit
* is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies beginning approximately 2 weeks prior to administration of the initial dose of trial drug, throughout the trial, until the posttrial visit
* consumes greater than 3 glasses of alcoholic beverages daily
* consumes greater than 6 servings of coffee, tea, cola, energy-drinks, or other caffeinated beverages per day.
* is currently a regular or recreational user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within approximately 3 months

Exclusion Criteria (Parts II and III):

* has a history of diabetic ketoacidosis in the last 6 months.
* has had one or more severe hypoglycemic episodes associated with hypoglycemic seizures, comas or unconsciousness within 2 weeks prior to dosing
* has used systemic (intravenous, oral, inhaled) glucocorticoids within 3 months of screening or is anticipated to require treatment with systemic glucocorticoids during study participation
* has a history of hypersensitivity to pharmacologic insulins or to any of the inactive ingredients in regular human insulin, or to any E. coli-derived drug product

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2014-11-26 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2016-07-29 (Actual)

PRIMARY OUTCOMES:
Number of participants who experienced an adverse event | Up to 30 days following last dose
Pharmacokinetic parameter: steady state plasma concentration (Css) | Part I: final 30 minutes of each infusion rate; Parts II and III: final 30 minutes of each interval
Pharmacokinetic parameter: area under the plasma concentration curve from time 0 to infinity (AUC [0 to infinity]) | Part I: 18 time points between predose and 600 minutes (min.); Part II: 19 time points between predose and 535 min.; Part III: 18 time points between predose and 415 min. following start of infusion
Pharmacokinetic parameter: clearance (CL) | Part I: final 30 minutes of each infusion rate; Parts II and III: final 30 minutes of each interval
Pharmacokinetic parameter: volume of distribution (Vd) | Part I: final 30 minutes of each infusion rate; Parts II and III: final 30 minutes of each interval
Pharmacokinetic parameter: plasma apparent terminal half-life | Part II: following 9 hour infusion; Part III: following 7 hour infusion
Pharmacodynamic parameter: steady-state glucose infusion-rate (GIR) in Part II | Part II: during the final 60 minutes of the infusion
Number of participants who discontinued study drug due to an adverse event | Part I: 1 day; Parts II and III: 9 days

SECONDARY OUTCOMES:
Number of participants with anti-drug antibody (ADA) formation | Up to 30 days following last dose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Krug AW, Visser SAG, Tsai K, Kandala B, Fancourt C, Thornton B, Morrow L, Kaarsholm NC, Bernstein HS, Stoch SA, Crutchlow M, Kelley DE, Iwamoto M. Clinical Evaluation of MK-2640: An Insulin Analog With Glucose-Responsive Properties. Clin Pharmacol Ther. 2019 Feb;105(2):417-425. doi: 10.1002/cpt.1215. Epub 2018 Sep 30. PMID 30125349